CLINICAL TRIAL: NCT03187808
Title: The Effect of Single Thoracic Manipulation Combined With Special Massage Technique on Mechanical Neck Pain: A Randomized Controlled Trial
Brief Title: Effects of Single Thoracic Manipulation and Special Massage Technique (RT Technique) on Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, RAWIPORN PITHAK, Principle Investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BNOJPH-KKU-RP-001
Record Dates: First submitted 2017-01-16; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Neck Pain
Keywords: Neck pain, Thoracic manipulation, special massage
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A is a group of performing single thoracic manipulation at zygapophyseal joint of T6-T7.
  Interventions: Other: Single thoracic manipulation
- Group B (Experimental): Group B is a group of performing single thoracic manipulation combined with special massage technique (RT technique).
  Interventions: Other: Single thoracic manipulation; Other: Special massage technique (RT technique)

INTERVENTIONS:
Other: Single thoracic manipulation — The subjects, who were randomly allocated to single thoracic manipulation group, will receive the single thoracic manipulation interventions directly to both sides of zygapophyseal joints of T6-T7. Each subject will be asked to lie on prone position on an experimental table. After that, the researcher will mark on both sides of zygapophyseal joints of T6-T7. Then, the subject will be instructed to take a deep inhalation and exhalation. During the exhalation, the therapist will perform the single thoracic manipulation (screw thrust technique) at zygapophyseal joints of T6-T7. If the audio pop is not heard during the first attempt, the therapist will ask the subject to reposition and repeat the technique. The procedure will be performed for maximum of 2 attempts and within 2 minutes.
Other: Special massage technique (RT technique) — The special massage technique or RT technique is a treatment that was developed by Puntumetakul and colleagues in 2013 (copyright registration number 314783). The subjects in this group will be asked to lie on side lying position with 90 degrees of hip flexion and 90 degrees of knee flexion. The researcher will perform the RT technique by press their thumb on the treatment lines beside the posterior vertebral line from level of inferior angle of scapula to the lowest rib for 5 seconds per point and 3 sets per treatment line (Figure 8). Total time of this procedure is approximately 2 minutes.
  Arms: Group B

SUMMARY:
This study aims to compare the immediate effects of using a single thoracic manipulation combined with special massage technique (RT technique) and single thoracic manipulation alone on pain level at rest, cervical range of motion, upper limb neurodynamic test, neck disability, and adverse effects in chronic mechanical neck pain patients.

DETAILED DESCRIPTION:
- The subjects will be recruited through posted advertisements, and announcements, to find the patients who meet the criteria of mechanical neck pain that is the pain provoked by sustained prolonged neck posture, neck movement or palpation of cervical musculature. The subjects will be screened by screening questionnaire, and then will be examined by a physiotherapist. All subjects will be required to sign an inform consent before participating to the study

- The sample size was calculated by using the averaged of pain level at rest after treatment from the single thoracic manipulation combined with special massage group and single thoracic manipulation group, after the preliminary procedure that will be conducted with ten subjects per each group. After that, the variance was calculated by using the equation σ2 = (n1-1)s12 + (n2-1)s22/(n1+n2)-2 and the result will be used for calculate the sample size. A drop out rate will be set as 20%. The effect size (∆), the significant level of lower than 0.05 (Zα(0.05) = 1.96) and a power of test at 90 percent (Zβ(0.2)=1.28) was used to calculate in the equation as follow: n/group = "2(Zα + Zβ)2σ2" /"∆2"

ELIGIBILITY:
Inclusion Criteria:

* They have neck pain on posterior neck or shoulder, which is the area from superior nuchal line to spinous process of 1st thoracic vertebrae, with mechanical characteristics consisting of the symptoms provoked by sustained prolonged neck posture, neck movement or palpation of cervical musculature (Martı´nez-Segura et al., 2006).
* They have symptoms for at least 3 months in duration.
* They have pain level at rest at least mild level (from 3 score or greater) measured by Visual Analog Scale (Jensen et al., 2003).
* They have a baseline Neck Disability Index (NDI) Thai version score of 10% or greater (Suvarnnato et al., 2013).

Exclusion Criteria:

The subjects will be excluded from current study if they have the following conditions including:

1. Cervical radiculopathy or myelopathy
2. History of whiplash injury within 6 weeks of examination
3. History of cervical surgery or thoracic surgery
4. History of cervical or thoracic injuries including fracture or dislocation
5. Fibromyalgia syndrome
6. The serious spinal conditions including spinal osteoporosis, spinal tuberculosis, and tumors
7. History of treated by spinal manipulation within 2 months before participating in the study
8. The diseases that are contra-indication to receive a spinal manipulation, such as hypertension, heart disease and meningitis
9. Pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain level at rest | Change from baseline at 3 weeks
  A Visual Analog Scale (VAS) will be used for recording level of pain at rest.

SECONDARY OUTCOMES:
Cervical Range of Motion (CROM) | Change from baseline at 3 weeks
  The Cervical Range of Motion (CROM) device (Performance Attainment Associates, USA) will be used to measure the cervical range of motion, including flexion, extension, lateral flexion and rotation.
Upper limb tension test 1 (ULTT1) | Change from baseline at 3 weeks
  The details of performing ULTT1 can be described as follow: the examiner will stand at side of tested limb with turn facing towards patient's head, and hold patient's one hand to control his or her thumb and fingers. Next, the examiner will use other hand to keep patient's shoulder in depression position to prevent the movement of shoulder girdle elevation during shoulder abduction. Then, the examiner will perform shoulder abduction with 110 degrees, forearm supination with the wrist and fingers extend, laterally rotation of shoulder, and elbow extension respectively. The last component of the test is the examiner asked patient turning their head to opposite side of tested arm. In current study, the researcher will measure the changing response of first sequence, that patient have a symptoms, to investigate that the intervention may affect the neural tension or not.
The Neck Disability Index Thai version (NDI-TH) | Change from baseline at 3 weeks
  The Neck Disability Index Thai version (NDI-TH) questionnaire (Appendix C), which is a reliable instrument to assess functional disability in neck pain patients with high internal consistency (ICC = 0.85) (Uthaikhup et al., 2011), will be used to assess the subjects' perceived disability level which can be show the impact of their neck pain to the daily living.
Adverse effects | Change from baseline at 3 weeks
  After the intervention is complete, the subjects will be asked about any symptoms that are the side effect occurring from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: RUNGTHIP PUNTUMETAKUL, Ph.D, Study Director — Faculty of Associated Medical Science, Khon Kaen University

IPD SHARING:
Plan to Share IPD: No
The participants' data and documents in this study will not be shared to other researchers.